CLINICAL TRIAL: NCT06850259
Title: A Comparative Crossover Study on the Safety, Efficacy, and Patient Reported Satisfaction of the PureWick™ System With an Established Comparator Overnight in the Home Setting for Incontinence in Adult Males
Brief Title: This Study Will Collect Clinical and Patient Reported Satisfaction Data From Males Requiring Urine Output Management Overnight in the Home Setting.
Acronym: PUREST-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UCC-24HC013
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Urinary Incontinence
Keywords: PureWick Urine Collection System; male external catheter; urinary incontinence; urine management; nocturia; nocturnal enuresis
MeSH Terms: conditions — Urinary Incontinence; Nocturia; Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Sequence 1 (Experimental): PureWick™ System is used first, followed by cross-over to UltraFlex™
  Interventions: Device: PureWick™ System; Device: UltraFlex™ Self-Adhering Male External Catheter
- Treatment Sequence 2 (Experimental): UltraFlex™ is used first, followed by cross-over to PureWick™ System
  Interventions: Device: PureWick™ System; Device: UltraFlex™ Self-Adhering Male External Catheter

INTERVENTIONS:
Device: PureWick™ System — The PureWick™ System consists of the PureWick™ Urine Collection System used with the PureWick™ Male External Catheter (MEC), which is intended for non-invasive urine output management in male patients. The PureWick™ MEC is a single-use, non-sterile, commercially available device, which is Class I, 510(K) exempt.
Device: UltraFlex™ Self-Adhering Male External Catheter — UltraFlex™ is a self-adhering male external catheter used for the drainage of urine. The catheter is applied by the patient or caregiver. The self-adhering male external catheter is designed for the management of adult male urinary incontinence.

SUMMARY:
This post-market study will assess the performance of and user satisfaction with the PureWick™ Male External Catheter in a home setting. The study will also observe safety of the study device and collect information from participants about their experience using the device.

DETAILED DESCRIPTION:
Approximately 15 men requiring the use of diapers or pads at night for urine management will take part in this prospective, open-label, crossover trial. Participants will be 1:1 randomized to a treatment sequence using two devices: the PureWick™ System (PureWick™ Male External Catheter & PureWick™ Urine Collection System) and the UltraFlex™ Self-Adhering Male External Catheter. Participants will use each urine management device overnight while sleeping for a period of 7 days with a 2-day washout period in between. Total duration of participation is approximately 16 days. The primary efficacy endpoint is the mean capture rate. The primary safety endpoint is the number of device-related AEs requiring medical intervention. Capture rates and Adverse Events are assessed daily throughout each 7-day treatment phase. Sleep disturbance is assessed at baseline and every 7 days during treatment. End of study preference questionnaire is completed at the end of treatment. Device adherence is assessed by the proportion of device wear nights that the study device became dislodged. Tolerability is assessed by number of nights of actual device use.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male participants ≥ 65 years of age at the time of signing the informed consent
2. Male anatomy at the time of enrollment
3. Currently use diapers, pads, or equivalent at night for urine output management
4. Willing to comply with all study procedures in this protocol
5. Provision of signed and dated informed consent form

Exclusion Criteria:

1. Has frequent episodes of bowel incontinence; or
2. Has chronic urinogenital infections, active genital herpes; or
3. Has Urinary retention; or
4. Has experience using study devices in the home setting within the last year; or
5. Is agitated, combative, and/or uncooperative and may remove the external catheter; or
6. Has any wound, open lesion or irritation on the genitalia, perineum, or sacrum; or
7. Any other condition that, in the opinion of the investigator, would preclude them from participating in the study; or
8. Is considered a vulnerable population.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Performance of the PureWick MEC in the Home Setting | Daily for 7 days during each treatment phase
  Capture rate following void (captured as % of urine captured by device and collected in canister, measured by weight).
  Prior to each nightly use, the weight of the empty urine collection canister and the weight of a dry absorbent pad are collected. Participants use the device overnight while sleeping with the absorbent pad underneath them. The next morning, the post-void weight of the urine collection canister and the post-void weight of the absorbent pad are collected.
  Capture rate is calculated as the weight of captured urine (post-void canister weight - pre-void canister weight) / total urine volume (captured urine (post-void canister weight - pre-void canister weight) + leaked urine (post-void pad weight - pre-void pad weight)) * 100.
Number of device-related Adverse events requiring medical intervention | Daily for 7 days during each treatment phase
  Number of device-related Adverse events requiring medical intervention, such as new prescription medication, surgery or procedure, or therapy ordered by a medical provider to treat or manage the adverse event, in each treatment group.

SECONDARY OUTCOMES:
Participant Device Preference | After completion of both 7-day treatment phase or at the time of treatment discontinuation, whichever comes first.
  Preference questionnaire administered after completion of both treatments to assess participant device satisfaction and preference for the PureWick MEC or UltraFlex sheath-style male external catheter. Participants will select which of the two devices they preferred and provide feedback on why the preferred device was selected.
Participant Device Tolerance | After completion of each 7-day treatment phase or at the time of treatment discontinuation, whichever comes first.
  Participant's tolerability is determined by the number of days of actual device use
Device Adherence/Dislodgement | After completion of each 7-day treatment phase or at the time of treatment discontinuation, whichever comes first.
  Proportion of device wear nights that each device became dislodged.

OTHER OUTCOMES:
Participant Sleep Quality | Starting at baseline and then after completion of each 7 day treatment phase.
  The PROMIS Sleep Disturbance Short Form 4a score collected at baseline and after each 7 day treatment phase. The PROMIS Sleep Disturbance 4a contains 4 scored items each scored from 1 to 5. All item raw scores are computed into a total score where higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Finlay Medical Research, Greenacres City, Florida
  - Trialfinity Clinical Research Center, Hamilton, New Jersey

IPD SHARING:
Plan to Share IPD: No